CLINICAL TRIAL: NCT02237976
Title: Interest of Learning Self-hypnosis in Patients Awaiting Lung Transplantation
Brief Title: Self-hypnosis in Patients Awaiting Lung Transplantation
Acronym: SelfHypTp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/47; 2014-A00538-39 (Other: ANSM)
Record Dates: First submitted 2014-09-09; First posted 2014-09-12 (Estimated); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Lung Transplantation
MeSH Terms: interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-hypnosis (Experimental): Patients are trained to practice self-hypnosis wen they are listed for lung transplantation. They are encourage to practice it before and after transplantation.
  Interventions: Behavioral: Self-hypnosis
- Routine practice (Active Comparator): No specific intervention
  Interventions: Behavioral: Routine practice

INTERVENTIONS:
Behavioral: Self-hypnosis
  Arms: Self-hypnosis
Behavioral: Routine practice
  Arms: Routine practice

SUMMARY:
The proposed study is designed to utilize a self-hypnosis training program for patients awaiting lung transplantation. This technique can increase their well being, particularly by decreasing postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 15 years or more requiring lung transplantation

Exclusion Criteria:

* patients who cannot participate in learning sessions of self-hypnosis for cultural , cognitive or environmental reasons
* patients who have participated in only one learning self-hypnosis session before transplantation

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2014-07-31 (Actual); Primary Completion 2017-04-26 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Pain after lung transplantation | one month
  Mean pain score in the 48 hours preceding the consultation performed one month after lung transplantation. Pain score is determined by the patient on a visual analogue scale (VAS) .

SECONDARY OUTCOMES:
Pain before and after lung transplantation | 6 months
  Pain score is determined by the patient on a visual analogue scale (VAS) at the time of inscription on waiting list for transplantation, at the 8th day post transplantation, one and four months after transplantation
Anxiety | 6 months
  Anxiety is determined by the patient on a visual analogue scale (VAS) at the time of inscription on waiting list for transplantation, at the 8th day post transplantation, one and four months after transplantation.
  Anxiety is also determined by
  * the State Anxiety Inventory and the Trait Anxiety Inventory at the time of inscription on waiting list for transplantation,
  * the State Anxiety Inventory one and four months after transplantation.
Coping | 6 months
  Coping is determined by the patient (Coping Strategies Questionnaire) at the time of inscription on waiting list for transplantation, and four months after transplantation
Catastrophism | 6 months
  Catastrophism is determined by the patient (Sullivan questionnaire) at the time of inscription on waiting list for transplantation, and four months after transplantation
Quality of life | 6 months
  Quality of life is determined by the patient (SF12 questionnaire) at the time of inscription on waiting list for transplantation, one and four months after transplantation
Quality of life related to the procedure | 6 months
  Quality of life related to the procedure is determined by the patient using a specific questionnaire (Ringsted et al. Pain-related impairment of daily activities after thoracic surgery: a questionnaire validation. The Clinical Journal of Pain 2013;29(9):791-799) four months after transplantation
Practice of self-hypnosis | 6 months
  Practice of self-hypnosis is determined by the patient using a specific questionnaire at the 8th day post transplantation, one and four months after transplantation.
Forced expiratory volume in one second | 6 months
  Forced expiratory volume in one second is measured 4 months after transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Mireille Michel-Cherqui, MD, Principal Investigator — Hopital Foch
Locations (1):
- Hôpital Foch, Suresnes, Hauts De Seine, France